CLINICAL TRIAL: NCT02087592
Title: Prospective Randomized Multicenter Trial to Assess the Feasibility of a Structured Physical Exercise Training and Mediterranean-style Diet in Women With BRCA1/2 Mutations
Brief Title: Feasibility of Lifestyle Intervention in BRCA1/2 Mutation Carriers
Acronym: LIBRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIBRE-F-110013
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Hereditary Breast and Ovarian Cancer
Keywords: hereditary breast and ovarian cancer (HBOC); BRCA1/2 mutation carriers; Mediterranean diet; Structured exercise training; prevention
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual standard of care
- Intervention (Experimental): Usual standard of care plus structured physical exercise training plus mediterranean-style diet
  Interventions: Behavioral: Structured exercise training plus mediterranean diet

INTERVENTIONS:
Behavioral: Structured exercise training plus mediterranean diet
  Arms: Intervention

SUMMARY:
BRCA1/2 mutation carriers have a considerably increased risk to develop breast and ovarian cancer during their lifetime. There is evidence from the literature that for sporadic breast cancer disease risk and the course of disease can be significantly influenced by physical activity, nutrition and weight. The hypothesis of this 3 year, prospective randomized multicenter feasibility trial is that a structured life-style intervention program with exercise training and mediterranean diet is feasible and improves the nutritional and fitness status as well as the weight, the quality of life and stress reacting capacity.

ELIGIBILITY:
Inclusion Criteria:

* women with proven pathogenic BRCA1/2 mutation

Exclusion Criteria:

* metastatic tumor disease
* life expectancy <3 years
* clinically limiting cardiovascular or respiratory disease
* significant orthopedic disability which prevents from participating in the exercise training
* severe concomitant disease which prevents from participating in the group interventions
* Karnofsky index <60
* VO2max >150%
* Maximal exercise capacity < 50 W
* food allergies which prevent from mediterranean diet
* vegan diet
* body mass index <15 kg/m2
* pregnancy
* insufficient knowledge of German language
* insufficient compliance
* active participation in other interventional trials
* no informed consent

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Number of patients successfully completing the intervention program | 3 months

SECONDARY OUTCOMES:
Stress coping capacity (TICS) | 3 months
Grade of optimism (LOT) | 3 months
Body mass index as a marker of caloric balance | 3 months
Total fat intake | 3 months
maximum exercise capacity (VO2max) as a marker of physical fitness | 3 months
Quality of life (SF-36) | 3 months
Physical activity (IPAQ questionnaire) | 3 months

OTHER OUTCOMES:
Anthropometric parameters (waist and hip circumference, skinfold measurements) | 3 months
Body composition (body impedance analysis) | 3 months
Eating behaviour | 3 months
Laboratory parameters | 3 months
Aerobic exercise capacity during ergometry | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marion Kiechle, Prof. Dr., Principal Investigator — Technical University of Munich; Martin Halle, Prof. Dr., Study Director — Technical University of Munich; Stephan C Bischoff, Prof. Dr., Study Director — Universitaet Hohenheim, Stuttgart; Wolf-Dieter Gerber, Prof. Dr., Study Director — Universitaetsklinikum Schleswig-Holstein, Campus Kiel; Markus Loeffler, Prof. Dr., Study Director — University of Leipzig; Christoph Engel, Dr., Study Director — University of Leipzig; Rita K Schmutzler, Prof. Dr., Study Director — University of Cologne; Alfons Meindl, Prof. Dr., Study Director — Technical University of Munich
Locations (3):
- Germany (3):
  - University of Cologne, Cologne
  - University of Schleswig-Holstein Campus Kiel, Kiel
  - Technische Universitaet Muenchen, Munich

REFERENCES:
- [Derived] Seethaler B, Neyrinck AM, Basrai M, Kiechle M, Delzenne NM, Bischoff SC. Elucidating the effect of the Mediterranean diet on fecal bile acids and their mediating role on biomarkers of intestinal barrier function: An exploratory analysis of a randomized controlled trial. Life Sci. 2025 Oct 15;379:123855. doi: 10.1016/j.lfs.2025.123855. Epub 2025 Jul 26. PMID 40721110
- [Derived] Seethaler B, Lehnert K, Yahiaoui-Doktor M, Basrai M, Vetter W, Kiechle M, Bischoff SC. Omega-3 polyunsaturated fatty acids improve intestinal barrier integrity-albeit to a lesser degree than short-chain fatty acids: an exploratory analysis of the randomized controlled LIBRE trial. Eur J Nutr. 2023 Oct;62(7):2779-2791. doi: 10.1007/s00394-023-03172-2. Epub 2023 Jun 15. PMID 37318580
- [Derived] Seethaler B, Nguyen NK, Basrai M, Kiechle M, Walter J, Delzenne NM, Bischoff SC. Short-chain fatty acids are key mediators of the favorable effects of the Mediterranean diet on intestinal barrier integrity: data from the randomized controlled LIBRE trial. Am J Clin Nutr. 2022 Oct 6;116(4):928-942. doi: 10.1093/ajcn/nqac175. PMID 36055959
- [Derived] Berling-Ernst A, Yahiaoui-Doktor M, Kiechle M, Engel C, Lammert J, Grill S, Dukatz R, Rhiem K, Baumann FT, Bischoff SC, Erickson N, Schmidt T, Niederberger U, Siniatchkin M, Halle M. Predictors of cardiopulmonary fitness in cancer-affected and -unaffected women with a pathogenic germline variant in the genes BRCA1/2 (LIBRE-1). Sci Rep. 2022 Feb 21;12(1):2907. doi: 10.1038/s41598-022-06913-1. PMID 35190584
- [Derived] Seethaler B, Basrai M, Vetter W, Lehnert K, Engel C, Siniatchkin M, Halle M, Kiechle M, Bischoff SC. Fatty acid profiles in erythrocyte membranes following the Mediterranean diet - data from a multicenter lifestyle intervention study in women with hereditary breast cancer (LIBRE). Clin Nutr. 2020 Aug;39(8):2389-2398. doi: 10.1016/j.clnu.2019.10.033. Epub 2019 Nov 2. PMID 31735538
- [Derived] Kiechle M, Dukatz R, Yahiaoui-Doktor M, Berling A, Basrai M, Staiger V, Niederberger U, Marter N, Lammert J, Grill S, Pfeifer K, Rhiem K, Schmutzler RK, Laudes M, Siniatchkin M, Halle M, Bischoff SC, Engel C. Feasibility of structured endurance training and Mediterranean diet in BRCA1 and BRCA2 mutation carriers - an interventional randomized controlled multicenter trial (LIBRE-1). BMC Cancer. 2017 Nov 10;17(1):752. doi: 10.1186/s12885-017-3732-4. PMID 29126396
- [Derived] Hebestreit K, Yahiaoui-Doktor M, Engel C, Vetter W, Siniatchkin M, Erickson N, Halle M, Kiechle M, Bischoff SC. Validation of the German version of the Mediterranean Diet Adherence Screener (MEDAS) questionnaire. BMC Cancer. 2017 May 18;17(1):341. doi: 10.1186/s12885-017-3337-y. PMID 28521737
- [Derived] Kiechle M, Engel C, Berling A, Hebestreit K, Bischoff S, Dukatz R, Gerber WD, Siniatchkin M, Pfeifer K, Grill S, Yahiaoui-Doktor M, Kirsch E, Niederberger U, Marter N, Enders U, Loffler M, Meindl A, Rhiem K, Schmutzler R, Erickson N, Halle M. Lifestyle intervention in BRCA1/2 mutation carriers: study protocol for a prospective, randomized, controlled clinical feasibility trial (LIBRE-1 study). Pilot Feasibility Stud. 2016 Dec 19;2:74. doi: 10.1186/s40814-016-0114-7. eCollection 2016. PMID 28031860